CLINICAL TRIAL: NCT07328750
Title: Dynamic Q Angle And Core Endurance In Adolescent Athletes With Patellofemoral Pain Syndrome: A Sex-Based Comparative Retrospective Study
Brief Title: Dynamic Q Angle and Core Endurance in Adolescent Athletes With Patellofemoral Pain Syndrome
Acronym: PFPS-QCORE
Status: Recruiting | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: TM-FLEX-BAL-2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Postural Balance; Athletic Performance
Keywords: Y-Balance Test; Trunk Mobility; Digital Inclinometer; Sports-Specific Biomechanics; Elite Male Athletes; Adolescent Sports Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Wrestling Athletes: Elite adolescent male wrestlers. No intervention is administered; participants undergo standardized clinical and biomechanical assessments including trunk mobility (digital inclinometer), hamstring flexibility (Straight Leg Raise), and functional balance (Y-Balance Test).
  Interventions: Other: Observational Clinical and Biomechanical Assessment
- Sprint Athletes: Elite adolescent male sprint runners. No intervention is administered; the same standardized assessment protocol is applied, including trunk mobility, hamstring flexibility, and Y-Balance Test performance.
  Interventions: Other: Observational Clinical and Biomechanical Assessment
- Canoe/Kayak Athletes: Elite adolescent male canoe/kayak athletes. No intervention is administered; participants complete the same biomechanical assessment battery as the other cohorts.
  Interventions: Other: Observational Clinical and Biomechanical Assessment
- Taekwondo Athletes: Elite adolescent male taekwondo athletes. No intervention is administered; all assessments are performed using the standardized trunk mobility, flexibility, and functional balance testing protocol.
  Interventions: Other: Observational Clinical and Biomechanical Assessment

INTERVENTIONS:
Other: Observational Clinical and Biomechanical Assessment — No intervention is administered in this study. Participants only undergo standardized observational assessments, including trunk mobility measurements using a digital inclinometer, hamstring flexibility testing with the Straight Leg Raise test, and functional balance evaluation using the Y-Balance Test. No therapeutic or experimental procedures are applied.
  Other Names: Standardized Functional Evaluation Protocol

SUMMARY:
This cross-sectional observational study aims to compare trunk mobility, lower extremity flexibility, and functional balance performance across different sports branches in adolescent elite male athletes. Trunk mobility will be assessed using a digital inclinometer in flexion, extension, and rotational movements; hamstring flexibility will be evaluated using the Straight Leg Raise test; and functional balance will be measured using the normalized Y-Balance Test. The study seeks to identify sport-specific biomechanical characteristics and potential indicators related to injury risk and performance adaptations in adolescent competitive athletes.

DETAILED DESCRIPTION:
Adolescent elite athletes are exposed to sport-specific mechanical loading patterns that may lead to adaptations in trunk mobility, flexibility, and dynamic balance control. These biomechanical characteristics may differ between sports branches due to variations in postural demands, training volume, movement strategies, and neuromuscular control mechanisms. Understanding inter-sport differences may contribute to performance optimization and preventive rehabilitation approaches in youth athletics.

This study is designed as a cross-sectional, observational, and multi-group comparative investigation including elite adolescent male athletes from different sports branches. All participants will undergo standardized clinical and biomechanical assessments. Trunk mobility will be measured using a digital inclinometer in flexion, extension, and rotation at the lumbosacral and thoracolumbar regions. Hamstring flexibility will be assessed using the passive Straight Leg Raise test, and functional balance will be evaluated using the Y-Balance Test composite score normalized to limb length.

The primary objective of the study is to compare functional balance performance across sports branches. Secondary objectives include comparing trunk mobility and hamstring flexibility measures and examining potential associations among these biomechanical parameters. The findings of this study are expected to provide evidence-based insight into sport-specific musculoskeletal characteristics and may support the development of targeted screening and injury-prevention strategies for adolescent elite athletes.

ELIGIBILITY:
Inclusion Criteria:

1. Male adolescent elite athletes aged 15-17 years
2. Licensed and actively training and competing in their respective sports branch
3. Minimum 3 years of continuous training experience
4. Ability to complete all clinical and biomechanical assessments
5. Written informed consent (parental consent for minors)

Exclusion Criteria:

1. Acute musculoskeletal injury within the past 3 months
2. Chronic lower extremity or spinal pathology
3. History of orthopedic surgery within the past 6 months
4. Neurological, metabolic, or systemic condition affecting movement or balance
5. Inability to comply with the testing protocol or incomplete data

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Elite adolescent male athletes aged 15-17 years from different sports branches (wrestling, sprint, canoe/kayak, and taekwondo). Participants are recruited from sports performance centers and evaluated using standardized trunk mobility, flexibility, and functional balance assessments.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Y-Balance Test Composite Score (%) | Baseline (single assessment at study enrollment)
  Dynamic functional balance performance assessed using the Y-Balance Test. Composite score is calculated from normalized anterior, posteromedial, and posterolateral reach distances on the dominant limb.

SECONDARY OUTCOMES:
Trunk Mobility - Inclinometer Range of Motion (°) | Baseline (single assessment at study enrollment)
  Spinal mobility measured using a digital inclinometer in flexion, extension, and rotation at the lumbosacral and thoracolumbar regions. Values are recorded in degrees on the dominant side.
Hamstring Flexibility - Straight Leg Raise Angle (°) | Baseline (single assessment at study enrollment)
  Passive Straight Leg Raise test performed on the dominant lower extremity using a goniometer. The maximum tolerated angle is recorded in degrees.
Body Composition (Descriptive Variable) | Baseline (single assessment at study enrollment)
  Body fat percentage
Body Composition (body mass index) | Baseline (single assessment at study enrollment)
  body mass index obtained using a multi-frequency bioelectrical impedance device (profiling purpose only; not included as a primary outcome).

CONTACTS AND LOCATIONS:
Overall Officials: burcin ugur tosun, Study Chair — Ministry of Youth and Sports, Olympic Preparation Center, Adana, Türkiye
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus